CLINICAL TRIAL: NCT03010085
Title: A Multicenter Randomized Controlled Trial of Open Versus Laparoscopic Left-sided Hepatectomy
Brief Title: Open Versus Laparoscopic Left-sided Hepatectomy Trial
Acronym: OLLEH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Collaborators: Korea Cancer Center Hospital (Other); Seoul National University Boramae Hospital (Other); Eulji University Hospital (Other); Bucheon St. Mary's Hospital (Other); Gyeongsang National University Hospital (Other); Jeju National University Hospital (Other); The Catholic University of Korea (Other); Soonchunhyang University Hospital (Other); Inje University (Other); Pusan National University Hospital (Other); DongGuk University (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Chonnam National University Hospital (Other); Hallym University Kangnam Sacred Heart Hospital (Other); Hallym University Medical Center (Other); Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Huisong Lee, Dr., Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OLLEH trial
Record Dates: First submitted 2016-11-30; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Neoplasm, Liver
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Open left-sided hepatectomy) (Active Comparator): Open left-sided hepatectomy Laparotomy (upper midline, inverted 'L', or Benz incision) Mobilization of the liver Glissonian approach or individual isolation technique Left lateral sectionectomy or left hemihepatectomy
  Interventions: Procedure: Open left-sided hepatectomy
- B (Laparoscopic left-sided hepatectomy) (Experimental): Trocar insertion Mobilization of the liver Glissonian approach or individual isolation technique Left lateral sectionectomy or left hemihepatectomy
  Interventions: Procedure: Laparoscopic left-sided hepatectomy

INTERVENTIONS:
Procedure: Open left-sided hepatectomy — Open left-sided hepatectomy Laparotomy (upper midline, inverted 'L', or Benz incision) Mobilization of the liver Glissonian approach or individual isolation technique Left lateral sectionectomy or left hemihepatectomy
  Other Names: Left-sided hepatectomy; Left lateral sectionectomy; Left hemihepatectomy
  Arms: A (Open left-sided hepatectomy)
Procedure: Laparoscopic left-sided hepatectomy — Trocar insertion Mobilization of the liver Glissonian approach or individual isolation technique Left lateral sectionectomy or left hemihepatectomy
  Other Names: Laparoscopic left lateral sectionectomy; Laparoscopic left hemihepatectomy
  Arms: B (Laparoscopic left-sided hepatectomy)

SUMMARY:
Open versus Laparoscopic Left-sided Hepatectomy (OLLEH) trial Multi-institutional, prospective and randomized trial in patients undergoing left sided hepatectomy through laparoscopic versus open procedure.

Primary endpoint: Functional recovery Secondary endpoint: Hospital duration, estimated blood loss, operation time, resection margin status, postoperative complication, mortality, liver function laboratory test, re-admission, quality of life, cosmesis, cost effectiveness

DETAILED DESCRIPTION:
Laparoscopic left-sided hepatectomy is widely performed for the treatment of various hepatic neoplasms. Many studies have reported that laparoscopic left-sided hepatectomy is safe and effective compared with open conventional left-sided hemihepatectomy. However, prospective study is rare and there is no randomized controlled trial.

The surgeons who are affiliated at a medical center in capital area of Korea launched the Open versus Laparoscopic Left-sided Hepatectomy (OLLEH) trial to verify the surgical outcome of laparoscopic left-sided hepatectomy.

Laparoscopic surgery has benefits that less wound and less pain. The hypothesis of the study is 'The laparoscopic left-sided hemihepatectomy is better than open surgery from functional recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who underwent open or laparoscopic left-sided hepatectomy for benign or malignant neoplasm of the liver
2. Child-Pugh A without portal hypertension

   * No portosystemic shunt
   * No splenomegaly
   * Platelet count >100,000/ul
3. Age 18 to 80
4. Eastern Cooperative Oncology Group performance status: 0 or 1
5. American society of anesthesiology class: I or II
6. Informed consent

Exclusion Criteria:

1. Additional intervention to the liver (Radio Frequent Ablation, Percutaneous Ethanol. Injection Therapy or others)
2. Combined hepatectomy
3. Bile duct reconstruction
4. Intrahepatic duct stone
5. Upper abdominal laparotomy history
6. Previous hepatectomy
7. Combined operation for extrahepatic disease
8. Vulnerable population (mental retardation, pregnancy)
9. Patient who participated in other clinical trial within 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Checklist of functional recovery (Questionnaire, liver function test of aspartate aminotransferase and alanine aminotransferase) | up to 30 days
  Checklist of functional recovery
  1. (Questionnaire) Do you want intravenous analgesics for postoperative pain ? (Yes, No)
  2. (Questionnaire) Do you have trouble to ambulate by oneself ? (Yes, No)
  3. (Questionnaire) Do you have trouble to digest solid meal ? (Yes, No)
  4. (Questionnaire) Do you want intravenous fluid to subside your thirsty ? (Yes, No)
  5. (Liver function test) Are serum aspartate aminotransferase and alanine aminotransferase increasing ? (Yes, No)
     * Daily check the five item above until every item is 'No'
     * If all of the items are 'No', the patient is regarded as a functionally recovered state.

SECONDARY OUTCOMES:
Postoperative complication | up to 30 days
  Discharge summary
Mortality | up to 30 days
  Death within 30 days after surgery
Readmission rate | up to 30 days
  Readmission
Hospital duration | up to 30 days
  Hospital duration after surgery
Blood loss | up to 30 days
  Estimated blood loss on anesthesiology sheet
Operation time | up to 30 days
  Skin incision to wound closure
Resection margin status | up to 30 days
  According to the pathology report
Liver function test | up to 30 days
  Bilirubin, Aspartate Aminotransferase, Alanine Aminotransferase, Prothrombin time, international normalized ratio (INR), Albumin
Quality of life | up to 30 days
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Electronic case report form — http://ollehkorea.com